CLINICAL TRIAL: NCT06980415
Title: Testing Children's Visual Acuity at Home: The Feasibility of a Home-based Visual Acuity Test to Improve Outcomes From Patching for Amblyopia.
Brief Title: Children's Eye Examination and Testing At Home Study
Acronym: CHEETAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RHM OPH0285
Record Dates: First submitted 2023-09-01; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2023-09

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Visual acuity test (Experimental)
  Interventions: Device: Kay Pictures iSight

INTERVENTIONS:
Device: Kay Pictures iSight — Tablet-based visual acuity measurement

SUMMARY:
Repeated measures observational study of tablet-based children's visual acuity tests.

DETAILED DESCRIPTION:
The most common disease seen in paediatric eye clinics is lazy eye (amblyopia), which affects 5% of the population. Amblyopia is treated using eye patching or eye drop therapy over the course of 6 months to two years. Up to half of all children undergoing therapy for amblyopia do not achieve a successful outcome. The outcome measure (visual acuity) is how small a letter the patient can see on a Snellen-like chart. Visual acuity is measured six-weekly for amblyopia patients in the outpatient clinic and is used to decide when to start therapy and how much therapy to use.

Recent developments by visual acuity test manufacturers of iPAD-based tests have simplified the testing protocol so that it may be performed by untrained staff. It is currently not understood to what level of accuracy a lay-person can perform the test. The present study was conceived to answer questions brought to us by patients and their parents, whom reported in our PPI activities that they feel they could use the iPAD themselves to test visual acuity.

This study is designed to quantify the correlation between iPAD-based visual acuity measurements taken by lay persons and the gold-standard, clinic-based measurements taken by qualified orthoptists using standard of care equipment and protocols. Collaboration between the PPI group and researchers expect that the correlation will likely be high and the teams anticipate possible advantages to lay-persons testing the visual acuity including, fewer visits to hospital and better adherence to amblyopia therapy.

Home visual acuity test has potential to reduce the number of outpatient clinic assessments or allow assessment of patients that could not be assessed during the UK coronavirus epidemic. However, the awarding body, BIOS, have requested that orthoptists do not instruct patients to use home-based visual acuity tests as the procedure is not covered by indemnity insurance. BIOS reference a lack of evidence-base. The new aim of the study will be to determine the validity of home-based visual acuity assessments with the possibility of providing such an evidence- base.

The study aim will be achieved by measuring the visual acuity in the outpatient clinic as per standard of care and asking the parent or carer to use the iPAD to test visual acuity at the same visit

ELIGIBILITY:
Inclusion Criteria:

* Age under 10 years
* Able to complete a subjective visual acuity test

Exclusion Criteria:

* Parent or carer not willing to participate in the study and give written informed consent

Ages: 0 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Visual acuity | Participants complete the primary outcome variable measurements on Day 0 of study recruitment.
  Visual acuity collected using the Kay Pictures iSight iPad application in the hands of the parent or carer on Day 0 of the study (cross sectional design).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD available upon request to Daniel Osborne (d.osborne@soton.ac.uk)